CLINICAL TRIAL: NCT06201130
Title: Airway Microbiome Changes After Artificial Airway Exchange in Critically-ill Pediatric Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-23-0420
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Tracheostomy; Endotracheal Tube; Ventilator Associated Pneumonia; Tracheitis; Microbial Colonization; Pediatric Infectious Disease; Pediatrics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Tracheitis; Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum aspirates from endotracheal tubes or tracheostomies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Suctioning of artificial airway — Collection of tracheal aspirates in either the PICU or NICU will occur. We will instill 1 mL of normal saline, then perform bag ventilation, and then suction out aspirate. Suctioning is routinely performed for tracheostomy and endotracheal tube hygiene - for instance, it is performed on tracheostomies by caregivers at home. The aspirates that will be collected will be clinically indicated and otherwise would be discarded. If the patients weren't enrolled in this research, the aspirates would have been collected anyways.

SUMMARY:
Artificial airways, such as endotracheal tubes and tracheostomies, in the pediatric and neonatal intensive care units (PICU, NICU respectively) are lifesaving for patients in respiratory failure, among other conditions. These devices are not without a risk of infection - ventilator-associated infections (VAIs), namely ventilator associated pneumonia (VAP) and ventilator-associated tracheitis (VAT), are common. Treatment of suspected VAI accounts for nearly half of all Pediatric Intensive Care Unit (PICU) antibiotic use. VAI can represent a continuum from tracheal colonization, progression to tracheobronchial inflammation, and then pneumonia. Colonization of these airways is common and bacterial growth does not necessarily indicate a clinically significant infection. Tracheostomies, which are artificial airways meant for chronic use, are routinely exchanged on a semi-monthly to monthly basis, in part to disrupt bacterial biofilm formation that aids bacterial colonization and perhaps infection. When patients with tracheostomies are admitted for acute on chronic respiratory failure or a concern for an infection, these artificial airways are also routinely exchanged at some institutions. There however remains a critical need to understand how an artificial airway exchange alters the bacterial environment of these patients in sickness and in health. This research hypothesizes that exchanging an artificial airway will alter the microbiome of the artificial airway, by altering the microbial diversity and relative abundance of different bacterial species of the artificial airway. This study will involve the prospective collection of tracheal aspirates from patients with artificial airways. We will screen and enroll all patients admitted to a the NICU or PICU at Cohen Children's Medical Center (CCMC) who have tracheostomies and obtain tracheal aspirates within 72 hours before and after tracheostomy or endotracheal tube exchange. Tracheal aspirates are routinely obtained in the NICU and PICU from suctioning of an artificial airway and is a minimal risk activity. These samples will be brought to the Feinstein Institutes for Medical Research for 16 s ribosomal DNA (16srDNA) sequencing, which allows for accurate and sensitive detection of relative abundance and classification of bacterial flora. Tracheal aspirate sets will be analyzed against each other. Additionally, clinical and epidemiological data from the electronic medical record will be obtained. Antibiotic exposure will be accounted for via previously published means.

ELIGIBILITY:
Inclusion Criteria:

* All patients with tracheostomies in the pediatric or neonatal intensive care unit
* Patients with endotracheal tubes undergoing artificial airway exchange in the pediatric or neonatal intensive care unit

Exclusion Criteria:

* None

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects included will be children aged 0-18 years of all sexes, ethnic and racial backgrounds. Subjects will generally be ill and have many comorbid conditions, as patients with artificial airways in the PICU and NICU tend to have complex issues. There are no exclusion criteria. Children must be included as this study wishes to understand the impact of exchanging artificial airways in the pediatric population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-06-26 (Estimated); Study Completion 2025-06-26 (Estimated)

PRIMARY OUTCOMES:
Shannon diversity index | December 2023-June 2025
  A measure of alpha diversity
Bray-curtis dissimilarity | December 2023-June 2025
  A measure of beta diversity
Differential abundance | December 2023-June 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Can share identified data

REFERENCES:
- [Background] Kuhl LP, Marostica PJC, Macedo AJ, Kuhl G, Siebert M, Manica D, Sekine L, Schweiger C. High microbiome variability in pediatric tracheostomy cannulas in patients with similar clinical characteristics. Braz J Otorhinolaryngol. 2023 Mar-Apr;89(2):254-263. doi: 10.1016/j.bjorl.2022.05.001. Epub 2022 May 20. PMID 35680554
- [Background] Maffei D, Brewer M, Codipilly C, Weinberger B, Schanler RJ. Early oral colostrum administration in preterm infants. J Perinatol. 2020 Feb;40(2):284-287. doi: 10.1038/s41372-019-0556-x. Epub 2019 Nov 20. PMID 31748654
- [Background] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Background] Perez-Losada M, Graham RJ, Coquillette M, Jafarey A, Castro-Nallar E, Aira M, Freishtat RJ, Mansbach JM. The temporal dynamics of the tracheal microbiome in tracheostomised patients with and without lower respiratory infections. PLoS One. 2017 Aug 10;12(8):e0182520. doi: 10.1371/journal.pone.0182520. eCollection 2017. PMID 28796800
- [Background] Perez-Losada M, Graham RJ, Coquillette M, Jafarey A, Castro-Nallar E, Aira M, Hoptay C, Freishtat RJ, Mansbach JM. Tracheal Microbiota in Patients With a Tracheostomy Before, During and After an Acute Respiratory Infection. Pediatr Infect Dis J. 2018 Nov;37(11):e269-e271. doi: 10.1097/INF.0000000000001952. PMID 29462107
- [Background] Zachariah P, Ryan C, Nadimpalli S, Coscia G, Kolb M, Smith H, Foca M, Saiman L, Planet PJ. Culture-Independent Analysis of Pediatric Bronchoalveolar Lavage Specimens. Ann Am Thorac Soc. 2018 Sep;15(9):1047-1056. doi: 10.1513/AnnalsATS.201802-146OC. PMID 29877714